CLINICAL TRIAL: NCT04492488
Title: An Open-Label, Multi-center Phase I/II Dose Escalation and Expansion Study to Assess the Safety, Efficacy and Pharmacokinetics of MRG002 in Patients with HER2-Positive Advanced Solid Tumors and Locally Advanced or Metastatic Gastric/Gastroesophageal Junction (GEJ) Cancer
Brief Title: A Study of MRG002 in Patients with HER2-Positive Advanced Solid Tumors and Locally Advanced or Metastatic Gastric/Gastroesophageal Junction (GEJ) Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRG002-101
Record Dates: First submitted 2020-07-23; First posted 2020-07-30 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumors; Advanced or Metastatic Gastric Cancer; Advanced or Metastatic Gastroesophageal Junction Cancer
Keywords: MRG002; Antibody Drug Conjugate (ADC); HER2; Solid tumors; Gastric/GEJ Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Solid Tumors (Experimental): Phase I Dose Escalation: MRG002 will be administrated by an IV infusion of escalating doses (starting dose of 2.2 mg/kg, followed by 2.6 mg/kg) on Day 1 of every 3 weeks (21-day cycle).
  Interventions: Drug: MRG002
- Locally Advanced or Metastatic Gastric/GEJ Cancer (Experimental): MRG002 will be administrated by an IV infusion on Day 1 of every 3 weeks (21-day cycle).
  Interventions: Drug: MRG002

INTERVENTIONS:
Drug: MRG002 — Administrated intravenously

SUMMARY:
The objective of this study is to assess the safety, efficacy, and pharmacokinetics of MRG002, as well as the immunogenicity as defined by the incidence of anti-drug antibody (ADA) of MRG002 in patients with HER2-positive advanced solid tumors and locally advanced or metastatic gastric/gastroesophageal junction (GEJ) cancer.

DETAILED DESCRIPTION:
This study consists of two parts. In Part A, patients will receive MRG002 as a monotherapy at doses of 2.2 or 2.6 mg/kg intravenously (IV) over 60-90 minute on Day 1 of every 3 weeks (Q3W), to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D). In part B, patients will receive a single IV infusion of MRG002 at RP2D on Day 1 of Q3W.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be able to provide written informed consent and follow the requirements specified in protocol.
* Age: ≥18 years.
* Life expectancy ≥6 months.
* Must have histologically or cytologically confirmed HER2-positive metastatic, unresectable cancer and must have had prior disease progression on all standard therapies for their tumor.
* Available archival tumor tissue (archival or from a new biopsy).
* At least one non-irradiated measurable tumor lesion according to RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Acceptable liver, renal, hematologic and coagulation function.

Exclusion Criteria:

* Toxicities (except alopecia & fatigue) due to prior antitumor therapy are higher than CTCAE v5.0 Grade 1.
* Toxicities due to radiotherapy (higher than grade 1) have not resolved to CTCAE v5.0 Grade ≤1 at least 21 days prior to the screening visit.
* Prior palliative or therapeutic radiation therapy to any RECIST v1.1 target lesion that defines baseline measurable disease for the study.
* Untreated or uncontrolled central nervous system (CNS) metastases.
* Any chemotherapy, biotherapy, immunotherapy, radiotherapy or other anti-tumor therapy within 3 weeks of the first dose of study treatment.
* Any severe cardiac dysfunction within 6 months of enrollment.
* Pulmonary embolism or deep vein thrombosis within 3 months prior to the first dose of study drug.
* Concurrent malignancy within 5 years prior to entry.
* Uncontrolled hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure > 100 mmHg).
* History of ventricular tachycardia, or torsade des pointes.
* History of moderate to severe dyspnea at rest due to advanced malignancies or their complications, severe primary lung disease, current need of continuous oxygen therapy, or clinically active interstitial lung disease (ILD) or pneumonitis.
* Major surgery within 4 weeks of the first dose of study treatment and not fully recovered. Minor surgery within 2 weeks prior to study treatment.
* Known allergic reactions to any component or excipient of MRG002 or known allergic reactions to trastuzumab or other prior anti-HER2 or other monoclonal antibody ≥ Grade 3.
* Patients who have any known liver disease, including chronic hepatitis B, hepatitis C, autoimmune hepatic disorders, primary biliary cirrhosis or sclerosing cholangitis; Patients who have concurrent, serious, uncontrolled infections or known infection with HIV, or have a diagnosed acquired immunodeficiency syndrome (AIDS); or an uncontrolled autoimmune disease, or have undergone organ transplant.
* Active uncontrolled bacterial, viral, fungal, rickettsial, or parasitic infection.
* Any severe and/or uncontrolled systemic disease that at the discretion of investigator and sponsor makes it undesirable for the patient to participate in this study.
* Use of systemic corticosteroids within 4 weeks prior to the first dose of treatment.
* Use of strong CYP3A4 inhibitors.
* Pregnancy or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | DLT will be evaluated during the first 21-day treatment cycle (Cycle 1)
  The dose level in which (i) less than 2 out of 6 patients in a treatment cohort experiences dose-limiting toxicity (DLT); or (ii) <33% of an evaluable patient treatment cohort experiences DLT.
Recommended Phase II Dose (RP2D) | Day 1 to Day 21 of Cycle 1
  Identify the recommended Phase II dose (RP2D) of MRG002 for Phase II clinical study. The RP2D may be the same as the MTD or an evaluable dose level lower than the MTD.
Objective Response Rate (ORR) | Baseline to study completion (24 months)
  Objective response rate (ORR) will be assessed by Independent Central Review (ICR) based on RECIST v1.1. Cumulative safety and dosing data will be reviewed by an independent Data Safety Monitoring Board (DSMB).
Incidence of Adverse Events (AEs) | After signing informed consent until 45 days after the last dose of MRG002
  AEs will be coded using MedDAR. Descriptive statistics will be used to summarize results to assess the safety and tolerability profile of MRG002.

SECONDARY OUTCOMES:
Duration of Response (DoR) | Baseline to study completion (24 months)
  Sensitivity analyses of DoR from the Investigator's assessment will be performed in the final analysis.
Disease Control Rate (DCR) | Baseline to study completion (24 months)
  Sensitivity analyses of DCR from the Investigator's assessment will be performed in the final analysis.
Progression Free Survival (PFS) | Baseline to study completion (24 months)
  Sensitivity analyses of PFS from the Investigator's assessment will be performed in the final analysis.
Pharmacokinetics (PK) parameter for MRG002: Maximum Drug Concentration (Cmax) | Baseline to study completion (24 months)
  Cmax will be derived from the PK blood samples collected and will be summarized with descriptive statistics.
PK parameter for MRG002: Area Under the Curve Up to the Last Validated Measurable Plasma Concentration (AUClast) | Baseline to study completion (24 months)
  AUClast will be derived from the PK blood samples collected and will be summarized with descriptive statistics.
PK parameter for total antibody (TAb): Cmax | Baseline to study completion (24 months)
  Cmax will be derived from the PK blood samples collected and will be summarized with descriptive statistics.
PK parameter for TAb: AUClast | Baseline to study completion (24 months)
  AUClast will be derived from the PK blood samples collected and will be summarized with descriptive statistics.
PK parameter for Monomethyl Auristatin E (MMAE): Cmax | Baseline to study completion (24 months)
  Cmax will be derived from the PK blood samples collected and will be summarized with descriptive statistics.
PK parameter for MMAE: AUClast | Baseline to study completion (24 months)
  AUClast will be derived from the PK blood samples collected and will be summarized with descriptive statistics.
Immunogenicity | Baseline to study completion (24 months)
  5 mL Blood samples for anti-drug antibody (ADA) analysis will be collected each time according to the pre-defined timepoints. The incidence of ADA will be summarized for all patients who received at least one administration of MRG002.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Denlinger, MD, Principal Investigator — Fox Chase Cancer Center
Locations (2):
- United States (2):
  - University of California Irvine Chao Family Comprehensive Cancer Center, Orange, California
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No